CLINICAL TRIAL: NCT05350540
Title: Randomized Phase II Study to Compare Intraoperative Indocyanine Green (ICG) Imaging and Guided Mucosal Debridement vs Observation (Standard of Care) to Reduce the Fistula Rate in Patients Undergoing Salvage Laryngectomy
Brief Title: Hypopharynx ICG to Reduce the Fistula Rate in Patients Undergoing Salvage Laryngectomy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Douglas Chepeha, MD, University Health Network, Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20-5419
Record Dates: First submitted 2022-04-15; First posted 2022-04-28 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Surgery Site Fistula

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICG (Experimental): This study will use intraoperative ICG imaging to assess recipient pharyngeal tissue perfusion. The ICG is the vascular contrast agent and the SPY Elite is the imaging device. 3mL of ICG will be injected using a peripheral IV access, followed by a 10mL saline flush. The pharyngeal mucosa will be imaged to quantify the tissue perfusion. Poorly perfused areas (less than 25%) will be debrided
  Interventions: Other: ICG dye
- Control (No Intervention): Patients assigned to the observation (control) group will undergo standard of care reconstruction of mucosa

INTERVENTIONS:
Other: ICG dye — Patients assigned to the intervention group will undergo surgery guided by tissue perfusion as directed by the ICG imaging
  Arms: ICG

SUMMARY:
A laryngectomy involves removing the voice box from the throat. After the voice box has been removed from the throat, the surgeon sews the throat closed. Sometimes part of the throat does not heal and saliva runs out of the throat. This is called a fistula. When a fistula happens, healing takes longer and patients will have to wait to eat and start speaking. The test in this research project is called ICG scan (indocyanine green) and tells the surgeon how much blood is flowing to different parts of the throat. If the test shows that there are parts of your throat that have low blood flow, which will delay healing. Only half of the patients in the study will get the ICG scan. This is so the patients who had the ICG scan can be compared to the patients that did not have the ICG scan to determine if the ICG scan really helps decrease fistulas.

DETAILED DESCRIPTION:
Salvage laryngectomy is associated with the highest morbidity and mortality in head and neck cancer patients. Pharyngocutaneous fistula is one of the most common surgical complication in the patient population and affects up to a third of patients undergoing total laryngectomy (TL) and pharyngolaryngectomy (PL). PCF is associated to increased rates of wound infections, prolonged hospitalization and vascular embarrassment (rupture and hemorrhage from major vessels). The use of vascularized flaps to assist in the reconstruction of the pharynx after laryngectomy have reduced the severity of complications patients experience after salvage laryngectomy. There is now interest in the quality of the vascular supply of the recipient pharyngeal tissue (pharyngeal mucosa). It is possible that vascular imaging of the recipient pharyngeal mucosa would provide the surgeon with intraoperative information that could guide pharyngeal mucosal debridement to remove any remaining pharyngeal tissue that has marginal vascularity (viability).

Initially developed in the 1950's, ICG imaging was used to assess retinal perfusion. Imaging acquisition with ICG uses a near-infrared wavelength (835nm) laser detection system. ICG imaging can also be used to direct debridement of marginally viable tissue. This approach has significantly reduced wound complications in patients undergoing breast reconstruction and colorectal surgery. ICG imaging has thus been found to be a reliable predictor of mucosal viability. Perfusion imaging studies in colorectal surgery, using laser fluorescence angiography, have shown a notable reduction in surgical revisions associated to anastomotic leaks, and a reduced hospitalization time. Preliminary reports in head and neck reconstructive surgery have shown an association between poor mucosal vascularity and higher fistula rate. In addition, ICG imaging and guided mucosal debridement suggest lower fistula rates.

We will be conducting a Phase II randomized trial study to assess the utility of ICG imaging for tissue perfusion, in order to reduce pharyngocutaneous fistula rate among patients undergoing salvage laryngectomy and vascularized tissue (flap) closure

ELIGIBILITY:
Inclusion Criteria:

* Signed written and voluntary informed consent.
* Patient must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other study procedures.
* Age > 18 years, male or female.
* Patient must be undergoing salvage laryngectomy after radiation or chemoradiation. By definition, the patients are considered resectable by the treating head and neck surgeon.
* The expected pharyngeal defect must be conducive to imaging with the ICG.
* Vascularized tissue augmentation (flap) is part of the operative plan (supra- or infraclavicular flap excludes the patient).
* ECOG performance status 0-2.

Exclusion Criteria:

* Total Laryngopharyngectomy
* On immune suppression medications
* Current hematologic malignancy
* Pregnancy
* Allergy to Iodine
* TSH greater than 8
* BMI less than 18
* Vascularized augmentation is a supra or infraclavicular rotational flap

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-11-11 (Actual); Primary Completion 2028-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
ICG Perfusion | Collected at time of surgery
  Perfusion of the mucosa after the administration of ICG will be recorded.
Surgical Complications | Collected up to 1 week after hospital discharge
  The complications the study participants experience post-surgically, if any, will be recorded.

SECONDARY OUTCOMES:
Disease Status | Collected at times week 1, 3 months, 6 months, and 12 months
  The health condition and disease stage of the participants will be collected at different time points.
Laryngeal Rehabilitation | Collected at times week 1, 3 months, 6 months, and 12 months
  Participants' means of communication using voice prosthesis or other devices will be collected at different time points.
Speech and Swallowing Questionnaire | Administered at times week 1, 3 months, 6 months, and 12 months
  This is a disease specific, 5-item, administered questionnaire to evaluate post-treatment speech and swallowing ability measure will provide critical data on the socialization of the patient as it relates to speaking and eating.

CONTACTS AND LOCATIONS:
Locations (1):
- University Health Network, Toronto, Ontario, Canada